CLINICAL TRIAL: NCT06636799
Title: EFFECTS OF MICRONEEDLING ON CLINICAL PARAMETERS OF STRIAE ALBA AND MORPHOLOGICAL PARAMETERS OF THE FEMALE TEGUMENTARY SYSTEM: A RANDOMIZED CLINICAL TRIAL
Brief Title: MICRONEEDLING ON CLINICAL PARAMETERS OF STRIAE ALBA AND MORPHOLOGICAL PARAMETERS OF THE FEMALE TEGUMENTARY SYSTEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabel de Almeida Paz (Other)
Responsible Party: Sponsor-Investigator, Isabel de Almeida Paz, MSc, University of the Sinos Valley
Organization: University of the Sinos Valley (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 6.584.696
Record Dates: First submitted 2024-09-20; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Striae; Atrophy
MeSH Terms: conditions — Striae Distensae; Atrophy | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Microneedling only (Experimental): In this procedure, only the derma roller composed of 1.5 mm microneedles from the Smart Derma Roller brand with 540 titanium needles was used.
  Interventions: Device: Microneedling only
- Microneedling associated with actives (Active Comparator): In this procedure, a derma roller composed of 1.5 mm microneedles from the Smart Derma Roller brand with 540 titanium needles associated with active ingredients were used.
  Interventions: Other: Microneedling and actives
- Control (No Intervention): This group did not receive intervention but participated in pre- and post-protocol assessments.

INTERVENTIONS:
Device: Microneedling only — In this procedure, a derma roller composed of 1.5 mm microneedles from the Smart Derma Roller brand with 540 titanium needles was used. The protocol was performed by passing the derma roller ten times in the following directions: horizontal, vertical, and diagonal right and left.
  Arms: Microneedling only
Other: Microneedling and actives — In this procedure, a derma roller composed of 1.5 mm microneedles from the Smart Derma Roller brand with 540 titanium needles was used. The protocol was performed by passing the derma roller ten times in the following directions: horizontal, vertical, and diagonal right and left. Group G3 received microneedling associated with active ingredients. This manipulated active ingredient was composed of growth factors (EGF Factor, TGFß3 Factor, and IDP-2 Peptide), Hydroxyprolisilane, and hyaluronic acid.
  Arms: Microneedling associated with actives

SUMMARY:
Stretch marks are dermal scars of multifactorial etiology, for which several treatments have been proposed. Among these is microneedling (MN), a technique that stimulates collagen production. However, the effects of MA alone and in combination with active agents on the length and area of stretch marks and the thickness of the integumentary system are not well understood, as the literature is scarce. Therefore, the objectives of this study were: To assess the effects of MA alone and in combination with active agents (growth factors, hyaluronic acid, and Hydroxyprolisilane CN®️) on clinical parameters (area and length) of stretch marks and morphological parameters (dermal and hypodermal thickness) of the female integumentary system. The sample was randomized into a control group (G1) that did not receive treatment, G2 that received MN alone, and G3 that received MN combined with active agents. Groups G2 and G3 underwent 3 sessions of the protocol with a 4-week interval. Groups were evaluated at the beginning and 4 months after the start of the protocol. Evaluation of the area and length of stretch marks was performed through photography, dermal and hypodermal thickness was assessed via ultrasonography, and satisfaction levels were measured using the Likert scale.

DETAILED DESCRIPTION:
This study was a randomized clinical trial in blocks with a 1:1 allocation, stratified by weight. The study was duly adapted to resolution 466/12 of the National Health Council on research involving human beings and to the Declaration of Helsinki. The evaluations and treatment protocols were carried out at the Physiotherapy Clinic of a Private Higher Education Institution.. The sample was characterized by convenience and healthy women who met the inclusion criteria were recruited, mainly via social networks. To calculate the sample size, the G-Power software (version 3.1.3; University of Trier, Trier, Germany) was used and the significance level adopted was α = 0.05 and power (1-β) = 0.80. No similar studies were found, so f 0.30 was used as the effect size. Therefore, the minimum number of participants required for the study was estimated at 24 participants. Considering possible losses during the protocol, 26 participants (+10%) were recruited. Randomization was performed by stratifying by weight. The randomization list was kept in opaque and sealed envelopes, ensuring that the allocation was hidden and random and that the therapist responsible for applying the microneedling had contact with the randomization only on the day of the protocol application. In the present study, the sample of 26 participants was divided into three groups. Group one (G1), control, composed of eight people, underwent all the evaluations, but did not receive the microneedling protocol or actives. Group two (G2), composed of nine people, underwent all the proposed evaluations and the isolated microneedling procedure. Group three (G3), composed of nine people, underwent all the proposed evaluations and the microneedling procedure associated with actives. Groups G2 and G3 underwent 3 sessions of the protocol with a 4-week interval. Groups were evaluated at the beginning and 4 months after the start of the protocol. Evaluation of the area and length of stretch marks was performed through photography, dermal and hypodermal thickness was assessed via ultrasonography, and satisfaction levels were measured using the Likert scale.This study adopted the intention-to-treat approach. Therefore, participants who did not attend the scheduled sessions were rescheduled, allowing all sessions planned to be carried out. When the decision was made to withdraw, the data collected up until the end were used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women (self-declaration of no diseases)
* Age between 18 and 35 years
* Presence of striae alba in the gluteal region

Exclusion Criteria:

* Health problems (cardiovascular, neurological, or musculoskeletal impairment)
* History of keloids
* Allergic disorders
* Skin cancer
* Systemic disease
* Diabetes mellitus
* Pregnant women
* Lactating women
* Psoriasis sufferers
* Hypersensitivity
* Use of peels, lasers, or any similar treatment in the last three months or any contraindication for performing microneedling.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The area of stretch marks | 30 minutes
  Photographic image analysis was performed before and after the protocol.These images will be analyzed later by tracing the area of the entire stria.
The thickness of stretch marks | 30 minutes
  Photographic image analysis was performed before and after the protocol. These images will be analyzed later by drawing a line between the upper and lower edges of the stria.

SECONDARY OUTCOMES:
Skin thickness | 30 minutes
  Ultrasound images collected before the first session and 30 days after the last session were analyzed. These images will be examined later, and the thickness of the skin will be evaluated.
Likert scale of patient satisfaction | 20 minutes
  A questionnaire was used to assess the level of satisfaction through non-standardized questions. Therefore, for adequate evaluation, in this study, patients undergoing microneedling post-treatment were asked about their level of satisfaction with the color, length and width of stretch marks, final skin quality, time of treatment and quality of care.
Hypodermis thickness | 30 minutes
  Ultrasound images collected before the first session and 30 days after the last session were analyzed. These images will be examined later, and the thickness of the hypodermis will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Paz, MSc, Principal Investigator — University of Vale dos Sinos
Locations (1):
- Universidade do Vale do Rio dos Sinos, São Leopoldo, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided